CLINICAL TRIAL: NCT02509910
Title: Implementation and Effects of Pulse-contour-automated SVV/CI Guided Goal Directed Fluid Therapy Algorithm for the Routine Management of Major Abdominal Surgery Patients
Brief Title: Implementation of a GDT Algorithm for Major Surgery Patients
Status: Completed | Type: Observational
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Dr. Thomas Kratz, MD, Philipps University Marburg
Other Study IDs: UKGMGDT
Record Dates: First submitted 2015-07-22; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Colectomy; Pancreatectomy; Fluid Therapy
Keywords: Major abdominal surgery; Goal directed therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard therapy: intraoperative standard fluid therapy for major abdominal surgery
- Goal directed therapy: intraoperative goal directed fluid therapy based on an angorithm lead by SVV/CI for major abdominal surgery patients

SUMMARY:
This study examines the effect of an algorithm for GDT for patients undergoing major surgery under routine conditions.

DETAILED DESCRIPTION:
Goal directed fluid management in major abdominal surgery has been shown to reduce perioperative complications. The approach aims to optimize the intravascular fluid volume by use of minimally invasive devices which calculate flow-directed variables such as stroke volume (SV) and stroke volume variation (SVV). The investigators aim to show the feasibility of routinely implementing such hemodynamic monitoring during major abdominal surgery, and to evaluate its effects in terms of perioperative fluid management and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* pancreatic surgery
* colorectal surgery

Exclusion Criteria:

* admission for revisional surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing major abdominal surgery (Colorectal and pancreatic surgery)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Length of stay in hospital | 90 days

SECONDARY OUTCOMES:
intraoperative crystalloid volume | 1 day
intraoperative colloid volume | 1 day
Length of stay at ICU | 90 days
Total amount of complications per patient | 90 days
Insufficiance of bowel anastomosis | 90 days
Pneumonia | 90 days
ACS | 90 days
acute renal failure | 90 days
Sepsis | 90 days
Intraabd. Infection | 90 days
wound infection | 90 days
UTI | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kratz, MD, Principal Investigator — Phillips University
Locations (1):
- University Hospital of Marburg, Department of Anesthesia, Marburg, Germany